CLINICAL TRIAL: NCT02006914
Title: Novel Therapy for Glucose Intolerance in HIV Disease
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Marie Gelato, Distinguished Service Professor, Stony Brook University
Other Study IDs: R21AT002499
Record Dates: First submitted 2011-08-11; First posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Insulin Resistance
Keywords: Insulin resistance; HIV disease; chromium picolinate
MeSH Terms: conditions — Insulin Resistance; Acquired Immunodeficiency Syndrome | interventions — picolinic acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fat and muscle biopsy samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Chromium Picolinate: Subjects who are HIV+ and insulin resistant
  Interventions: Dietary Supplement: Chromium Picolinate
- Placebo: HIV+ and insulin resistant

INTERVENTIONS:
Dietary Supplement: Chromium Picolinate — Subjects will be asked to take chromium picolinate; 2 tablets per day, 1000 mcg or a placebo for a total of 8 weeks.
  Other Names: Chromax
  Groups: Chromium Picolinate

SUMMARY:
This research is to investigate the nutritional supplement chromium picolinate. The investigators are testing to see how effective this supplement is in treating insulin resistance associated with HIV disease.

DETAILED DESCRIPTION:
This study will test the hypothesis that chromium picolinate improves insulin-stimulated glucose uptake by increasing the insulin receptor-mediated tyrosine phosphorylation of insulin receptor substrate-1, resulting in increased association with phosphatidylinositol 3-kinase.

Specific Aim 1 will assess quantitative improvements in insulin-mediated glucose disposal in a placebo-controlled clinical trial of chromium supplementation with 1000mpg (19.2 pmol) of chromium as chromium picolinate, overa two-month course of therapy. The investigators have shown that the insulin resistance (i.e. the inability of insulin to stimulate glucose uptake into peripheral tissues like muscle) in patients with HIV disease is associated with a defect in the insulin-signaling pathway leading from the insulin receptor, through phosphatidylinositol 3-kinase(PI 3-K, Figure 5). A similar defect in intracellular signaling has also been reported in patients with type 2 diabetes mellitus ):15-171. The cellular mechanism of improved insulin sensitivity with chromium supplementation will be determined in Specific Aim 2.

Specific Aim 2 will assess the effect of chromium supplementation on the insulin-stimulated activity of insulin receptor substrate-I-associated phosphatidylinositol 3-kinase in biopsies of muscle and fat tissue. This aim will also test the hypothesis that these physiological effects of chromium are mediated by alterations in the activity of insulin signaling. Understanding this mechanism may facilitate the design of even more effective strategies for improving insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and a diagnosis of HIV+ andlor AlDS made by standard CDC criteria.

Exclusion Criteria:

1. positive pregnancy test (all women must have a negative pregnancy test before beginning protocol);
2. diagnosis of cancer;
3. acute illness of any sort, however, patients may be enrolled once they are stable;
4. hemoglobin less than 11.0 gldl or hemodynamically unstable;
5. creatinine greater than or equal to 1.5 mgldl;
6. liver dysfunction as evidenced by elevations in transaminases 2-fold higher than upper limit of normal;
7. use of certain medications within the past month (e.g., glucocorticoids).
8. untreated hypertension (systolic BP > 150 mmHG, diastolic BP>100 mmHG);
9. patients with diabetes mellitus
10. hypogonadism
11. abnormal thyroid function (serum T'4 < 4 or > 12; TSH < 0.35 or > 5.5)
12. hepatitis C infection (if patients have had prior therapy and are now stable with no evidence of active infection they will be included. This will depend upon documentation from primary care giver).
13. CD4 counts below 300
14. viral load greater than 35,000.

Exclusion criteria (13) and (14) are added because the protocol requires that subjects be on a stable anti-retroviral regime for 3 months prior to study and 2 months on study. These criteria will make it less likely that anti-retroviral therapies will be switched in this subject population who are doing well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anyone with a positive diagnosis of HIV disease.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2005-06; Primary Completion 2010-05 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Chromium Picolinate supplementation | 8 weeks
  Hypothesis that chromium picolinate improved insulin-stimulated glucose uptake by increasing the insulin receptor-mediated tyrosine phosphorylation of insulin receptor substrate-1, resulting in increased association with phosphatidylinositol 3-kinase. There was a significant negative correlation between the fasting glucose levels and the insulin sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Marie C Gelato, MD, PhD, Principal Investigator — Stony Brook University School of Medicine Dept. Of Medicine/Endocrinology
Locations (1):
- Stony Brook University Hospital GCRC, Stony Brook, New York, United States

REFERENCES:
- [Result] Stein SA, Mc Nurlan M, Phillips BT, Messina C, Mynarcik D, Gelato M. Chromium Therapy for Insulin Resistance Associated with HIV-Disease. J AIDS Clin Res. 2013 Sep 7;4(9):239. doi: 10.4172/2155-6113.1000239. PMID 25346863